CLINICAL TRIAL: NCT04437342
Title: Postpartum Depression in the Covid-19 Pandemic and the Impact of Anaesthesia
Status: Completed | Type: Observational
Sponsor: General and Maternity Hospital of Athens Elena Venizelou (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Alexandra Hospital, Athens, Greece (Other); University of Ioannina (Other); Larissa University Hospital (Other)
Responsible Party: Principal Investigator, GEORGIA MICHA, Anaesthesiologist, MD, MSc, PhD, General and Maternity Hospital of Athens Elena Venizelou
Other Study IDs: Covid-19 Postpartum depression
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-10

CONDITIONS: Postpartum Depression; Psychological Stress; Maternal Distress
Keywords: postpartum depression; Covid-19 pandemic; anaesthesia
MeSH Terms: conditions — Depression, Postpartum; Stress, Psychological; COVID-19 | interventions — Patient Health Questionnaire; Weights and Measures; Psychiatric Status Rating Scales

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maternal Group: Pregnant women in labour (vaginal delivery or caesarean section) that are admitted to the hospital. Pre-labour 3 different questionnaires are administered to evaluate depression, general anxiety disorder and the association to the covid-19 pandemic. 40 days post delivery via telephone contact 2 questionnaires are administered, one in order to assess the postpartum disorder the other to assess depression.
  Interventions: Other: PHQ-9 (Patient Health Questionnaire) Depression Scale; Other: GAD-7 (General Anxiety Disorder) scale; Other: 38 questions questionnaire; Other: EPDS (Edinburgh Postnatal Depression Scale)

INTERVENTIONS:
Other: PHQ-9 (Patient Health Questionnaire) Depression Scale — 9 question questionnaire for assessment of depression
Other: GAD-7 (General Anxiety Disorder) scale — 7 question questionnaire for assessment of General Anxiety Disorder
Other: 38 questions questionnaire — 38 questions questionnaire
Other: EPDS (Edinburgh Postnatal Depression Scale) — 10 questions scale for detection of postpartum depression

SUMMARY:
The aim of this multicenter prospective study is to evaluate the association between the Covid-19 pandemic maternal psychological distress with the postpartum depression, demographic and anaesthesiologic variables

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women over the age of 18 that present for labour (vaginal delivery or caesarean section)

Exclusion Criteria:

* Not eligible in writing and reading in Greek
* Drug abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Maternity
Study Population: Pregnant women admitted to the hospital for vaginal delivery or caesarean section
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Correlation between the Covid-19 pandemic and postpartum depression with EPDS scale (Edinburgh postnatal depression scale) | 40 days postpartum
  Prevalence of postpartum depression during the Covid-19 pandemic with EPDS scale (Edinburgh postnatal depression scale)

SECONDARY OUTCOMES:
Correlation between the Covid-19 pandemic, postpartum depression and type of anaesthesia (general, epidural, spinal, combined, epidural analgesia for vaginal delivery) | 10 minutes postpartum
  Association between the Covid-19 pandemic, postpartum depression and type of anaesthesia (general, epidural, spinal, combined, epidural analgesia for vaginal delivery)
Correlation between the Covid-19 pandemic, postpartum depression and postpartum pain | 2 minutes prior to discharge from the Postanaesthesia care unit
  Association between the Covid-19 pandemic, postpartum depression and postpartum pain assessed during postanesthesia care unit stay assessed by Numeric Pain Rating Scale (Scale 0-10 where 0 equals no pain and 10 maximum possible pain)
Correlation between the Covid-19 pandemic, postpartum depression and postpartum pain | 2 minutes after admission to the Postanaesthesia care unit
  Association between the Covid-19 pandemic, postpartum depression and postpartum pain assessed during postanesthesia care unit stay assessed by Numeric Pain Rating Scale (Scale 0-10 where 0 equals no pain and 10 maximum possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Micha, PhD, Principal Investigator — Elena Venizelou General and Maternity Hospital of Athens, Greece
Locations (6):
- Greece (6):
  - "Elena Venizelou" General and Maternity Hospital of Athens, Athens, Attica
  - Aretaieio University Hospital, Athens, Attica
  - Alexandra Genaral Hospital Athens, Athens
  - University of Ioannina Health Science, Ioannina
  - University of Ioannina, Medical School, Ioannina
  - University of Thessaly Medical School, Larissa

IPD SHARING:
Plan to Share IPD: Yes
Research data, study protocol and statistical analysis plan will be available to the scientific community after publication. The corresponding author is responsible for reviewing these requests.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication of the article for indefinite time